CLINICAL TRIAL: NCT01249365
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK-580299) in Healthy Female Control Subjects From the Primary NCT00294047 Study
Brief Title: The Safety Evaluation of the GSK-580299 Vaccine in Women From the Control Group in the Primary NCT00294047 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113618; 2010-020227-48 (EudraCT Number)
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Infections, Papillomavirus
Keywords: medically significant conditions; cervical neoplasia; serious adverse events (SAEs); HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV vaccine (Experimental): Healthy female subjects aged 26 years and above, who received control vaccine in the primary study NCT00294047, were administrated 3 intramuscular injections of Cervarix vaccine into the deltoid of the non-dominant arm, according to a 0, 1, 6-month schedule in the current study.
  Interventions: Biological: GSK580299 (Cervarix)

INTERVENTIONS:
Biological: GSK580299 (Cervarix) — 3-dose schedule intramuscularly vaccination

SUMMARY:
This extension study is designed to assess the safety of GSK Biological's HPV vaccine GSK580299 in female subjects who took part in the primary study NCT00294047 and received the control vaccine in countries for which the licensed GSK HPV vaccine is not indicated for the subject's age group (26 years and older). This study is thus conducted to enable all women who received the control placebo in the primary NCT00294047 study to receive the GSK580299 vaccine.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, December 2010, leading to the update of 1 of the primary outcome measures and following Protocol Amendment 2, January 2011, leading to the removal of one of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* A subject previously enrolled in the study NCT00294047, who received the control vaccine, and who cannot receive the GSK580299 vaccine because the subject is above the age for which the vaccine is licensed.
* Written informed consent obtained from the subject
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or breastfeeding.
* A women planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase of the study, i.e. up to two months after the last vaccine dose.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen in the protocol.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days (i.e., Day 0-29) of each dose of vaccine, with the exception of administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine. Enrolment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

NOTE: Subjects enrolled in this study may also be eligible for a four-year gynaecological follow-up of the HPV-015 study, in which no investigational product will be administered. Subjects will be invited to the gynaecological follow-up study if either of the following applies:

* if they test positive for oncogenic HPV infection, but display normal cervical cytology at their concluding HPV-015 study end visit;
* if they are pregnant so that no cervical sample can be taken at their concluding HPV-015 study end visit;

  * Previous administration of any components of the vaccine.
  * Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
  * Cancer or autoimmune disease under treatment.
  * Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
  * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
  * History of any neurological disorders or seizures.
  * Acute disease and/or fever at the time of enrolment.
  * Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Australia (2):
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Portugal (5):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Setúbal
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Vaccine
Started | 199
Completed | 198
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | HPV Vaccine
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 1
  Geographic ancestry: Asian - Central/South Asian Heritage | 2
  Geographic ancestry: Asian - East Asian Heritage | 2
  Geographic ancestry: Asian - South East Asian Heritage | 78
  Geographic ancestry: White - Caucasian/European Heritage | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as the occurrence of any SAE regardless of intensity grade or relation to vaccination. Grade 3 SAE = SAE which prevented normal, everyday activities (in adults/adolescents, such an SAE, for example, prevented attendance at work/school and necessitated the administration of corrective therapy). Related SAE = SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the study (from Month 0 to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Vaccine
Number analyzed (Participants) | 199
Participants
  Any SAE(s) | 6
  Grade 3 SAE(s) | 2
  Related SAE(s) | 0

2. Primary Outcome: Number of Subjects Reporting Medically Significant Conditions (MSCs) and Potential Immune-mediated Diseases (pIMDs)
Description: Medically significant conditions (MSCs) are defined as:
  AEs prompting emergency room or physician visits that were not related to common diseases, or not related to routine visits for physical examination or vaccination; SAEs that were not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
  Potential immune-mediated diseases (pIMDs) are a subset of medically significant conditions that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
  Any was defined as the occurrence of any MSC or pIMD regardless of intensity grade or relation to vaccination. Grade 3 MSC or pIMD = a MSC or pIMD which prevented normal, everyday activities. Related MSC or pIMD = a MSC or pIMD assessed by the investigator as related to the vaccination.
Time Frame: Throughout the study (from Month 0 to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Vaccine
Number analyzed (Participants) | 199
Participants
  Any MSCs | 16
  Grade 3 MSCs | 2
  Related MSCs | 0
  Any pIMDs | 1
  Grade 3 pIMDs | 0
  Related pIMDs | 0

3. Primary Outcome: Number of Subjects Reporting Pregnancies and Outcome of Reported Pregnancies
Description: Live infant NO apparent congenital anomaly; Live infant congenital anomaly; Premature live infant NO apparent congenital anomaly; Premature live infant congenital anomaly; Elective termination NO apparent congenital anomaly; Elective termination congenital anomaly; Therapeutic abortion; Ectopic pregnancy; Spontaneous abortion NO apparent congenital anomaly; Spontaneous abortion congenital anomaly; Stillbirth NO apparent congenital anomaly; Stillbirth congenital anomaly; Molar pregnancy; Pregnancy ongoing; Lost to follow up.
Time Frame: Throughout the study (from Month 0 to Month 12)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered and who reported any pregnancies and outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Vaccine
Number analyzed (Participants) | 1
Participants
  Live infant NO apparent congenital anomaly | 1
  Live infant congenital anomaly | 0
  Premature live infant NO apparent congen. anomaly | 0
  Premature live infant congenital anomaly | 0
  Elective termination NO apparent congen. anomaly | 0
  Elective termination congenital anomaly | 0
  Therapeutic abortion | 0
  Ectopic pregnancy | 0
  Spontaneous abortion NO apparent congen. anomaly | 0
  Spontaneous abortion congenital anomaly | 0
  Stillbirth NO apparent congenital anomaly | 0
  Stillbirth congenital anomaly | 0
  Molar pregnancy | 0
  Pregnancy ongoing | 0
  Lost to follow up | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from the first receipt of study vaccine (Month 0) until 6 months following administration of the last dose of study vaccine (i.e. at study conclusion, Month 12).
Description: Non-serious solicited adverse events were not collected in this study. Non-serious unsolicited events collected in this study did not exceed the threshold of 5%.
Arm/Group | HPV Vaccine
All-Cause Mortality (participants affected / at risk) | 0/199
Serious Adverse Events (participants affected / at risk) | 6/199
Other Adverse Events (participants affected / at risk) | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV Vaccine (N=199)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1)
Agitated depression (Psychiatric disorders) | 1 (2)
Major depression (Psychiatric disorders) | 1 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.